CLINICAL TRIAL: NCT02235415
Title: Observation of the Efficacy and Tolerance of Motens® (Lacidipine) in Patients With Essential Hypertension, Under Normal Conditions Compared With an Open Clinical Trial
Brief Title: Observation of the Efficacy and Tolerance of Motens® (Lacidipine) in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 231.340
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — lacidipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Motens
  Interventions: Drug: Motens® (lacidipine)

INTERVENTIONS:
Drug: Motens® (lacidipine)

SUMMARY:
Study of the efficacy and tolerance of Motens® (lacidipine) in patients with essential hypertension. To obtain information on the dosage used in practice and the tolerance at the start of treatment (12 weeks)

ELIGIBILITY:
Inclusion Criteria:

Non-hospitalised patients of both sexes aged 18 years or more with essential hypertension requiring treatment according to the recommendations of the German League for Hypertension

Exclusion Criteria:

Patients who had the contraindications listed in the product information (the case report file contained a copy of the product information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential Hypertension recruited by General practicioners, cardiologists and specialists in internal medicine in non-Hospital practice
Sampling Method: Probability Sample
Enrollment: 24526 (Actual)
Dates: Start 1998-06; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy by the investigator on a 4-point verbal rating scale based on changes in blood pressure | Up to 12 weeks after start of drug administration
Assessment of tolerability by investigator on a 4-point verbal rating scale | Up to 12 weeks after start of drug administration
Number of patients with adverse events | Up to 12 weeks after start of drug administration